CLINICAL TRIAL: NCT04286061
Title: Efficacy of a Physiotherapy Intervention Through the Mobilization of Soft Tissues Assisted by Instruments in the Improvement of Mobility and Hip Strength in Semi-professional Rugby Players. A Randomized Clinical Study
Brief Title: Instrument-assisted Soft Tissue Mobilization to Improve Mobility and Hip Strength in Semi-professional Rugby Players
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Lockdown
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IASTM
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Rugby Player
Keywords: Rugby; Pubalgia; Strength; Range of motion; Instrument-assisted soft tissue mobilization.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each session will last 1 or 2 minutes, with one intervention being carried out a week, over a period of 4 weeks. Prior to the start of training, the instrument-assisted soft tissue mobilization technique will be performed
  Interventions: Other: Assisted soft tissue mobilization
- Control group (No Intervention): Players included in the control group will follow their usual training routine.

INTERVENTIONS:
Other: Assisted soft tissue mobilization — It will be done for 60 seconds, making a total of 30 strokes with the tool in the longitudinal direction to the muscle fibers. The physiotherapist will previously apply some massage cream to the area to be treated (adductor musculature) so that the tool slides at a 45º angle. Landslides will be made from the femoral condyle to the groin, and vice versa, exerting a pressure with the instrument of 3 over 10 on the analog visual scale that the subject feels
  Other Names: Experimental group
  Arms: Experimental group

SUMMARY:
Instrument-assisted soft tissue mobilization is a method that uses different devices to approach the myofascial system in variables such as joint mobility and muscle strength.

The objective of the study is to assess the effectiveness of the technique of soft tissue mobilization assisted by instruments in increasing the mobility of hip abduction and strength of the hip adductor musculature, in semi-professional rugby players federated in Spain of 18 at 32 years old Randomized, simple blind clinical study. 29 rugby players will be randomized to the two study groups: experimental (assisted soft tissue mobilization in the adductor leg muscles) and control (without intervention). The intervention will last 4 weeks, with 1 session per week, approximately 1 or 2 minutes each. The study variables will be hip abduction mobility (goniometry) and the strength of the hip adductor musculature (sphygmomanometry). A descriptive statistical analysis will be carried out calculating the main statistical characteristics. The distribution of normality will be calculated through an analysis of Saphiro Wilk. With the t-student test of repeated measures the differences will be calculated after the evaluations, and through an ANOVA of repeated measures the intra and intersubject effect will be calculated. The effect size will be calculated using the Cohen mean difference formula It is expected to observe an increase in hip abduction, as well as an increase in the strength of the adductor musculature of the hip.

ELIGIBILITY:
Inclusion Criteria:

* Male rugby players
* With an age range of 18 to 32 years
* Semi-professionals federated in Spain (category Division of Honor B, group C)
* Who have not had previous injuries to the lower limb in the last 2 months.

Exclusion Criteria:

* Subjects who: present any type of sensory alteration in the skin
* Are taking muscle relaxants
* Have skin infections
* Are allergic to the material of the intervention or evaluation tool
* Have not signed the informed consent document.

Ages: 18 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline range of motion of hip abduction after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  A long arm goniometer will be used, following the protocol described by Nussbaumer et al. . Before collecting the data, participants will perform a 5-minute warm-up on an exercise bike. The athlete will be placed supine, attached to the stretcher with a pelvic girth, with the contralateral leg hanging by the edge of the stretcher. The fixed arm of the goniometer will be placed on the transverse line formed by the superior antero iliac spines and the mobile arm on the longitudinal axis of the thigh, matching the goniometer fulcrum with the superior anterior iliac iliac spine of the lower limb to be evaluated. With the help of another physiotherapist, a passive and complete hip abduction will be performed, and the evaluator, in charge of the goniometer, will take the measurement resulting from the test.

SECONDARY OUTCOMES:
Change from baseline strength of the hip adductor muscle after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be assessed with a sphygmomanometer. The unit of measure will be millimeters of mercury (mmHg). The athlete will be placed in lateral recumbency with the leg to be evaluated extended and in contact with the stretcher and the contralateral leg at 90º of hip and knee flexion. The athlete will grab with his upper hand to the side of the stretcher and on his lower arm will support his head. The evaluator will place the pressure cuff (folded in thirds and preinflated to 10 mmHg) 5 cm proximally over the medial malleolus and secure it with a cinch that surrounds the stretcher. The athlete will exert a maximum isometric force against the pressure cuff and the webbing for 5 seconds. The test will be repeated 4 times, with a 30 second rest period between repetitions. The highest value of the 4 measurements will be chosen. A higher sphygmomanometer score will indicate greater strength of the hip adductor musculature (25,27).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided